CLINICAL TRIAL: NCT02766361
Title: Cognitive-Behavioral Rehabilitation Versus Treatment as Usual for Bipolar Patients
Brief Title: Cognitive-Behavioral Rehabilitation for Bipolar Disorder
Acronym: REHABBipolar
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Bernardo Carramão Gomes, PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNPQ 458144/2014-2
Record Dates: First submitted 2016-05-02; First posted 2016-05-09 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Psychotherapy; Cognitive rehabilitation
MeSH Terms: conditions — Bipolar Disorder | interventions — Cognitive Training; Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Rehabilitation (Experimental): 12 sessions of new intervention of cognitive behavior therapy and cognitive rehabilitation
  Interventions: Behavioral: Cognitive Behavioral Rehabilitation
- Treatment as Usual (Active Comparator): standard out-patient treatment offered in our clinic, which involves psychopharmacological mood stabilization and regular contacts with mental health nurses.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Rehabilitation — 12 weekly sessions of Combined intervention lasting 90 minutes
  Other Names: Combined intervention of CBT and Cognitive Rehabilitation
  Arms: Cognitive Behavioral Rehabilitation
Other: Treatment as Usual — standard out-patient treatment offered in our clinic, which involves psychopharmacological mood stabilization and regular contacts with mental health nurses.
  Arms: Treatment as Usual

SUMMARY:
The study consists of a clinical trial comparing a new structured group intervention, denominated "Cognitive-Behavioral Rehabilitation", to treatment as usual (TAU) for bipolar patients. The new approach is a combination of cognitive behavioral strategies and cognitive rehabilitation exercises, consisting of twelve weekly group sessions of 90 minutes each. To be included in the study, patients must be diagnosed with bipolar disorder, type I or II, be 18 to 55 years old, in full or partial remission and have an IQ of at least 80. A comprehensive neuropsychological battery, followed by mood, social functioning and quality of life assessments will occur in three moments: pre and post-intervention and after 12 months.

DETAILED DESCRIPTION:
Methods/Design The study compares Cognitive Behavioral Rehabilitation with Treatment as Usual (TAU), the latter being the commonly offered pharmacological treatment to bipolar patients. The psychological intervention will consist of twelve weekly group sessions, lasting 90 minutes each, and including 8 to 10 individuals. Subjects will be randomly assigned to one of the two arms, and submitted to a 12-month follow-up. During the entire study, all patients will be medicated accordingly to their clinical needs, and all changes in medication will be recorded as a secondary outcome , following the Necessary Clinical Adjustment (NCA) instrument. The NCA records medication adjustments implemented to reduce symptoms, improve response and functioning, or handle unbearable side effects.

Participants In order to be included, patients must be between 18 to 55 years old, literate, present an IQ score higher than 80 and have been diagnosed with bipolar I or II accordingly to DSM-V criteria (APA, 2014). Excluding conditions are: presence of substance or alcohol abuse in the last 6 months, current suicide risk, organic mental disorders or scores higher than 12, in the Montgomery-Asberg Depression Rating Scale (MADRS) or the Young Mania Rating Scale (YMRS) at the beginning of the interventions.

Recruiting will take place at an outpatient service provided by the Bipolar Disorder Research Program (PROMAN) at the University of São Paulo Medical School, Brazil. Patients will receive invitations individually, and sign an informed consent.

Procedure and Outcomes Once included, patients will complete the Portuguese versions of the following self-report questionnaires: the abbreviated instrument of quality of life (WHOQOL-bref), the Barratt Impulsiveness Scale 11 (BIS 11), the Social Skills Inventory (IHS) and the Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) . Patients will also complete the Functioning Assessment Short Test (FAST) and a brief questionnaire about bipolar disorder.

A brief neuropsychological battery will be conducted, which includes the Wechsler Abbreviated Scale of Intelligence (WASI) (Wechsler, 1999), and following subtests from the Cambridge Neuropsychological Test Automated Battery (CANTAB): Motor Screening Task (MOT); Rapid Visual Information Processing (RVP); Reaction Time (RTI); Spatial Span (SSP); Spatial Working Memory (SWM); One Touch Stockings of Cambridge (OTS); Pattern Recognition Memory (PRM); Delayed Matching to Sample (DMS); Attention Switching Task (AST); Emotion Recognition Task (ERT).

Subjects will also complete the initial assessment and mood module of the Structured Clinical Interview for DSM-5 (SCID-5) (APA, 2014) post-intervention at week 12, and 6 and 12 months thereafter.

Hypothesis

The study hypothesizes that Cognitive Behavioral Rehabilitation, in comparison to TAU, will:

I. Decrease the recurrence rates of new episodes; our primary outcome measure. II. Improve attention, mental flexibility, working memory and emotional recognition; our secondary outcome.

In an exploratory analysis we will also assess whether Cognitive Behavioral Rehabilitation may:

A. Enhances functional, social skills and quality of life scores; B. Increases sleep quality and knowledge about the disorder; and C., Reduces impulsivity

Interventions

Treatment as Usual (TAU) The control group from this study will receive standard out-patient treatment offered in our clinic, which involves psychopharmacological mood stabilization and regular contacts with mental health nurses. The number and amount of pharmacological treatment will follow the physician decision, respecting individual demands. All pharmacological treatment will be monitored and recorded in accordance to the Litmus study (Nierenberg et al. 2009).

Cognitive Behavioral Rehabilitation

We developed a 12-session intervention combining previous experience in cognitive behavior therapy for bipolar patients with several elements of cognitive remediation. The first step was to identify behaviors that have an important role in patients´ autonomy, followed by determining which cognitive domains are involved. The core objective was to promote the generalization of the learnt behaviors in the daily routine. Described below is the arrangement of each session, divided in three major Modules:

In the first Module comprises four sessions that attempt to improve attention and memory, considering the necessity to retain the information discussed throughout the sessions. There are two target behaviors involved: adherence to pharmacological treatment and mood monitoring. The cognitive remediation exercises seek to enhance verbal and visual memories, while secondarily enhancing attention with the paper material included in the manual. In the first session, group members and psychotherapists introduce themselves, followed by a discussion regarding the manual, individual´s expectations and the importance of attendance. The second session explores the concept of attention, and its importance as a door to further cognitive functions; the group also learns exercises aimed at training attention and memory. The third session focuses on medication adherence and its relation to attention. The core of the third session is the organization of the patient´s environment, which is frequently chaotic; a discussion about cues is encouraged at the end of the session. The fourth session starts by introducing mood graphics to patients and the importance of the early identifying of mood episodes. At the end of the first module, patients are stimulated to cook as method of reinforcing what they have learned while enhancing their autonomy.

The second module targets social cognition and communication. The fifth session familiarizes the patients with the concept of automatic thoughts (Rush and Beck, 1978), and a guide to identify its presence. Cognitive distortions are discussed along with examples provided by the subjects´ own experiences. The sixth session begins returning to the initial theme by habituating patients to the automatic thought record (Beck, 1997), patients are stimulated to restructure their own thoughts during experiences identified in previous sessions. Mental flexibility and empathy are introduced and discussed. The seventh session acquaint patients to assertive communication and emotion recognition by teaching role-playing exercises and the importance of positive assertiveness. The eighth session follows the same agenda as the seventh.

The last module of Cognitive Behavioral Rehabilitation aims at problem solving strategies and relapse prevention. The ninth session begins with the identification of personal problems, mainly by distinguishing it from preoccupations; the topic is important because patients often incorporate their problems to expectations and desires, generating an urge to abandon them, the session ends by emphasizing the importance of mental flexibility in generating as many responses as possible to each identified problem. In the tenth session, patients learn solving-problem techniques in a systematic setting. The eleventh session devotes to review information and clarify possible doubts from the patients; patients are also encouraged to debate the importance of regular routines and regular sleep, which can be adjusted using sleep hygiene techniques. A progressive muscle relaxation ends the session. Finally, the last session´s target is to avoid future mood relapses, it by returning to the personal goals defined in session one and prompting patients to develop a prevention plan. The acronym H.U.M.O.R. resumes the core points of the post-intervention maintenance program: 1) Habituate to a regular routine; 2) Use what you have learnt; 3) Monitor your mood; 4) Observe arising problems and deal effectively with it; and 5) Respond to automatic thoughts. All patients in the cognitive behavioral rehabilitation group will also receive TAU.

Statistical Analysis Sample Size The sample size calculation was based on the proportion of patients that remain episode-free after 12 months following a group intervention. Previous studies utilizing TAU exhibited a decrease of bipolar relapses in 30% of patients after a one-year follow-up. The present study anticipates a 55% success rate in prevention of mood relapses, during the same period, in patients assigned to the Cognitive Behavioral Rehabilitation. Thus, considering an 80% power to obtain a 5% significance, an estimated sample of 28 individuals per group, 56 in total, should be sufficient to achieve significant results. A previous study conducted by the same research team measured a drop-out rate of 10% in a one year follow-up, for this latter reason, the study will consist of 60 participants.

Baseline and Follow up Data. In order to measure the effects of the interventions, the study will employ the following statistical tests: 1) Qui-squared and Mann-Whitney to test homogeneity between the groups at the beginning of the interventions; 2) Student t test or Mann-Whitney to investigate the effects of such interventions, pre and post treatment, depending on the distribution of the data; 3) An analysis of variance, with and without adjustment for mood symptoms scores, IQ and BD duration, for comparison between groups; and 4) The Kaplan-Meyer survival method with log rank test for statistical analysis, to investigate the survival data between groups, which measures in weeks, the time to the first episode as an event.

ELIGIBILITY:
Inclusion Criteria:

* IQ higher than 80
* Bipolar I or II diagnoses
* Being literate

Exclusion Criteria:

* substance or alcohol abuse in the last 6 months,
* current suicide risk,
* organic mental disorders
* scores higher than 12, in the Montgomery-Åsberg Depression Rating Scale (MADRS) or the Young Mania Rating Scale (YMRS) at the beginning of the interventions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2020-11 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Interval to first mood episode | 6 months after the beginning of intervention group
  Survival data

SECONDARY OUTCOMES:
Change in Quality of life scores score WHOQOL | 3, 6 and 12 months after the beginning of intervention group
Change in Functionality Scale for Bipolar disorder (FAST) | 3, 6 and 12 months after the beginning of intervention group
Change in Barratt Impulsivity scale (BIS) | 3, 6 and 12 months after the beginning of intervention group
Change in Brian Sleep Scale | 3, 6 and 12 months after the beginning of intervention group
Change in Social skills scale (IHS) | 3, 6 and 12 months after the beginning of intervention group
Change in Motor Screening Task | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Rapid Visual Information Processing | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Reaction time Time Reaction time | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Spatial Span | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Spatial Working Memory | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in One Touch Stockings of Cambridge Change in Stockings of Cambridge | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Pattern Recognition Memory | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Delayed Change in Delayed Matching to Sample | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Change in Attention Switching Task | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST
Emotion Recognition Change in Emotion Recognition Task | 3, 6 and 12 months after the beginning of intervention group
  CANTAB SUBTEST

OTHER OUTCOMES:
Change in YMRS | 3, 6 and 12 months after the beginning of intervention group
  Young Mania Rating Scale
Change in MADRS | 3, 6 and 12 months after the beginning of intervention group
  Montgomery-Åsberg Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Beny Lafer, Professor, Principal Investigator — University of São Paulo Medical School, São Paulo, Brazil
Locations (1):
- Bipolar Disorder Program (PROMAN), Department of Psychiatry, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gomes BC, Rocca CC, Belizario GO, Lafer B. Cognitive-behavioral rehabilitation vs. treatment as usual for bipolar patients: study protocol for a randomized controlled trial. Trials. 2017 Mar 28;18(1):142. doi: 10.1186/s13063-017-1896-5. PMID 28351410